CLINICAL TRIAL: NCT05848635
Title: Hydromorphone for Perioperative Analgesia in Lung Tumor Ablation Parallel Controlled ：A Randomized, Parallel Controlled Trial
Brief Title: Hydromorphone for Perioperative Analgesia in Lung Tumor Ablation Parallel Controlled
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20221209
Record Dates: First submitted 2023-04-09; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Nodule; Ablation
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Lung tumor ablation using hydromorphone for pain control and anaesthesia (Experimental): Premedication:hydromorphone is started 15min before surgery with a single subcutaneous injection of 2mg.
  Intraoperative administration:NRS（Numeric Rating Scale）≥7 during operation, 2mg hydromorphone is injected intravenously and slowly pushed for 2-3 minutes.
  Postoperative administration:The drug is administered as needed according to the patient's postoperative pain, 2mg/time.
  Interventions: Drug: Hydromorphone Hydrochloride
- Active Comparator:Lung tumor ablation using morphine for pain control and anaesthesia (Active Comparator): Premedication:morphine is started 15min before surgery with a single subcutaneous injection of 10mg.
  Intraoperative administration:NRS（Numeric Rating Scale）≥7 during operation, 10mg morphine is injected intravenously and slowly pushed for 2-3 minutes.
  Postoperative administration:The drug is administered as needed according to the patient's postoperative pain, 10mg/time.
  Interventions: Drug: Morphine hydrochloride

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride — Drug: Hydromorphone Hydrochloride Hydromorphone hydrochloride injection is used for perioperative lung tumor ablation
  Other Names: Lung tumor ablation using hydromorphone hydrochloride
  Arms: Experimental: Lung tumor ablation using hydromorphone for pain control and anaesthesia
Drug: Morphine hydrochloride — Drug: Morphine Hydrochloride Morphine hydrochloride injection is used for perioperative lung tumor ablation
  Other Names: Lung tumor ablation using morphine hydrochloride
  Arms: Active Comparator:Lung tumor ablation using morphine for pain control and anaesthesia

SUMMARY:
This randomized, parallel controlled, single blind trial is designed to evaluate the efficacy and safety of hydromorphone versus morphine for perioperative analgesia in lung tumor ablation.

DETAILED DESCRIPTION:
Although the consensus of relevant guidelines and clinical studies recommend the use of opioids for perioperative analgesia in pulmonary tumor ablation surgery, there is a lack of specific analgesic programs for clinical reference. In view of the advantages of clinical application of hydromorphone and the lack of evidence for its application in perioperative analgesia of pulmonary tumor ablation, this study aims to explore the efficacy and safety of hydromorphone in perioperative analgesia of pulmonary tumor ablation, and provide some reference and suggestions for perioperative analgesia of pulmonary tumor ablation.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily attend and sign the informed consent form in person;
* Patients undergoing selective pulmonary tumor ablation;
* The Eastern Collaborative Oncology Group (ECOG) defines an activity status score of 2 or less;
* The estimated survival time is more than 3 months;
* Age 18-80, both sexes.

Exclusion Criteria:

* Severe coagulation dysfunction that cannot be corrected;
* History of severe cardio-cerebrovascular and respiratory diseases;
* Patients allergic to test drugs or contrast media;
* Patients with opioid addiction;
* Patients with cognitive dysfunction;
* Participated in other clinical investigators within three months;
* Investigators or their family members directly involved in the trial;
* Those who are deemed unfit to participate in the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Analgesic efficiency | The analgesia is evaluated at 1 hour before surgery, 5 minutes after the beginning of ablation
  effective cases / total cases * 100%. The NRS（Numeric Rating Scale） score ≤3 at all evaluation time points is considered as effective analgesia.

SECONDARY OUTCOMES:
Incidence of adverse reactions | perioperative period
  cases of adverse reactions / total cases * 100%

CONTACTS AND LOCATIONS:
Overall Officials: Xin Ye, graduate, Study Director — head of intervention department